CLINICAL TRIAL: NCT06203418
Title: Investigation of Multi-Family Therapy for Anorexia Nervosa
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Blue Cross Blue Shield (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0217
Record Dates: First submitted 2023-07-18; First posted 2024-01-12 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-05

CONDITIONS: Anorexia Nervosa
Keywords: Multi-Family Therapy
MeSH Terms: conditions — Anorexia Nervosa | interventions — Psychotherapy, Group

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Multi-Family Therapy
  Interventions: Behavioral: Multi-Family Therapy

INTERVENTIONS:
Behavioral: Multi-Family Therapy — Multi family therapy for anorexia nervosa (MFT-AN) draws on the same principles as FBT but is delivered in a more intensive format to help families to overcome a sense of isolation and stigmatization and to maximize their own resources. In the case of eating disorders, this program utilizes FBT principles (both approaches are guided by the family-based treatment philosophy, which stresses the impact of ED on family functioning and attempts to mobilize families as the primary agents of change in achieving recovery), and also utilizes learning from structural, systemic, strategic, narrative, and psychodrama-based family therapy practices,(Knatz et al., 2015). Generally between 5-7 families take part in MFT, sharing their experiences, learning by example, and providing support for one another. Study will utilize virtual adaptation of manualized treatment published by Simic et al 2021

SUMMARY:
The proposed project is an intensive multi family therapy (MFT) intervention involving patients with anorexia nervosa and their families. MFT interventions are informed from the principles of the family based treatment (FBT)/family therapy for Anorexia Nervosa (FT-AN) models. This program will offer families in vivo/virtual support while connecting with other families to increase knowledge of eating disorders and develop skills related to successfully supporting their adolescent during difficult times, including meal support and affect regulation. Our objective is to explore the influence of the MFT intervention on the primary outcome measures in eating disorder treatment, including weight, expressed emotion and eating disorder symptomatology.

DETAILED DESCRIPTION:
The proposed project is an intensive multi family therapy (MFT) intervention involving patients with anorexia nervosa and their families. MFT interventions are informed from the principles of the family based treatment (FBT)/family therapy for Anorexia Nervosa (FT-AN) models. This program will offer families in vivo/virtual support while connecting with other families to increase knowledge of eating disorders and develop skills related to successfully supporting their adolescent during difficult times, including meal support and affect regulation. Our objective is to explore the influence of the MFT intervention on the primary outcome measures in eating disorder treatment, including weight, expressed emotion and eating disorder symptomatology.

Families/patients will participate in an initial phone screen with the study coordinator to determine eligibility for the MFT. When participants are deemed eligible, they will then follow-up with a trained study assessor, where they will be consented for the study and complete both written and interview based assessments. Parents are welcome to participate without their child if their child does not wish to assent; the child may assent and participate in further treatment days if they wish. Families attending the group will continue to complete assessments throughout the study. Parents will complete the assessment interviews to their best knowledge about their child if their child does not choose to participate. Once a child agrees to participate, they will complete assessment interviews themselves. Patients will receive medical clearance/assessment by their primary care doctor or Eating Disorder medical provider prior to the start of the group. All medical assessments will be reviewed by Dr. Karen Bernstein. When "in person" group gatherings may resume, each treatment group will consist of 3-8 families with a new cohort starting approximately every 6 weeks (total of 6-8 sessions over a 1 year time period).

Accepted families will then by the 4 day MFT. Day 1 will involve a two hour orientation to the group. Families will learn the medical consequences of eating disorders, psychological principles of the treatment intervention, the expectations of participation, meet the treatment team, as well as hear from a family who has been through treatment. On the rest of day 1 through day 4, families will participate in a variety of planned activities aimed at facilitating change throughout the treatment process. Additionally, the "in person" group will have 3 3-6 hour follow up group sessions scheduled at 2 weeks post intervention (virtual), 1 month post intervention (in person), and 3 months post intervention (in person). In the virtual model, each treatment group will consist of 3-8 families with a new cohort starting approximately every 4-6 weeks (total of 8 -13 sessions over a 1 year time period). Day 1 will be a similar orientation as described above using the Zoom virtual platform. On the rest of day 1 and through day 4, families will participate in synchronous and asynchronous activities modified for the virtual format. Families in the virtual group will also participate in 3 3-hour follow up sessions in 2 weeks, 1 month, 3 months (all virtual).

Per the Multi-Family Therapy for Anorexia Nervosa Treatment Manual (Draft) (Simic M, Baudinet J et al), mechanisms of change in the group involve:

1. Multiple sources of input (parents, carers, young people, professionals) working together will allow participants to be both givers and receivers of new ideas/thoughts. Additionally, this will allow families to experiment with new behavioral interventions. The group is aimed at offering young people and their families the opportunity to experience simultaneous different roles. This process allows for new learning and experimentation with new ideas around the illness and family. Meeting families that are confronted with the same illness yet at different stages of recovery, makes experience sharing particularly rich and can inspire hope for change.
2. The MFT is designed purposefully with increased intensity and broadening of the treatment scope. Families receive a large dose of the treatment in the format of 4, 6 hour days (in person), or 4, 4 hour days with additional asynchronous tasks (virtual). The dose of treatment is created to match the intensity of the illness and promote behavioral experimentation and change within a short period of time. This 4 day "burst" has the primary aim of increasing parental efficacy in taking charge of the patient's illness. Families will participate in additional follow up sessions to "boost" and monitor the effects of the intervention
3. The MFT is designed to increase solidarity, reduce isolation, and facilitate building a community around behavioral change.

The overall themes of the intervention are engagement and understanding of the illness and its impact on the family, managing mealtimes and providing in vivo support during meals and process/problem solving around mealtimes, exploration of the impact of the illness of family relationships and working to set a path to improve them, and planning for the future (Simic M, Baudinet J et al). The intervention will include educational/cognitive behavioral, motivational, and problem-solving components, along with relational elements.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* living at home with at least one parent/guardian
* diagnosis of restricting eating disorder
* 11-18 years of age
* Medically stable per medical clearance form

Exclusion Criteria:

* Active psychosis (parent or child)
* Current dependence on drug or alcohol (parent or child)
* Past history/current abuse (sexual/physical), neglect

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-05-21 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Effect on Eating Disorder Symptomatology (multiple variables) - 1. weight | 1 year
  weight in lbs over time
Effect on Eating Disorder Symptomatology (multiple variables) - 2. BMI | 1 year
  BMI (kg/m^2): weight and height will be converted into appropriate units for calculation
Effect on Eating Disorder Symptomatology (multiple variables) - 3. Heart rate | 1 year
  Heart Rate (beats per minute)
Effect on Eating Disorder Symptomatology (multiple variables) - 4. eating disorder thoughts and behaviors | 1 year
  This is measured by 3 assessments that share scales. These assessments are the Eating Disorder Examination, Eating Disorder Examination Questionnaire and the Parent Eating Disorder Examination Questionnaire. Each of these measures have a total of 5 scales. These include Restraint, Eating Concern, Shape Concern and Weight Concern as well as a Global (total) score. This measured on a scale from 0-6 with 0 suggestion no presence of symptom and 6 representing maximum score. (Restraint, Eating Concern, Shape Concern and Weight Concern) and an overall global score, with a higher score indicating more problematic eating difficulties. Scale: 0-6
Effect on Eating Disorder Symptomatology (multiple variables) - 5. co-morbid psychiatric disorders | 1 year
  Co-morbid psychiatric disorders measured by Mini-International Neuropsychiatric Interview for Children and Adolescents (MiniKid) is a short standardized diagnostic interview and covers a rather broad range of diagnoses applicable to children and adolescents. This results in a 0 or 1 score. 0 of diagnosis is not given, 1 if diagnosis is given
Effect on Eating Disorder Symptomatology (multiple variables) - 6. co-morbid psychiatric disorders | 1 year
  Revised Children's Anxiety and Depression Scale (RCADS) is a 47-item, youth self-report questionnaire with subscales including: separation anxiety disorder, social phobia, generalized anxiety disorder, panic disorder, obsessive compulsive disorder, and low mood (major depressive disorder). It also yields a Total Anxiety Scale (sum of the 5 anxiety subscales) and a Total Internalizing Scale (sum of all 6 subscales). To score the RCADS manually, each item is assigned a numerical value from 0-3, where 0 = Never, 1 = Sometimes, 2 = Often, and 3 = Always. Higher number suggests higher severity.
Effect on Eating Disorder Symptomatology (multiple variables) - 7. co-morbid psychiatric disorders | 1 year
  Hospital Anxiety and Depression Scale (HADS) Hospital Anxiety and Depression Scale (HADS) - Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression.
  is a 47-item, youth self-report questionnaire with subscales including: separation anxiety disorder, social phobia, generalized anxiety disorder, panic disorder, obsessive compulsive disorder, and low mood (major depressive disorder). It also yields a Total Anxiety Scale (sum of the 5 anxiety subscales) and a Total Internalizing Scale (sum of all 6 subscales). To score the RCADS manually, each item is assigned a numerical value from 0-3, where 0 = Never, 1 = Sometimes, 2 = Often, and 3 = Always. Higher number suggests higher severity.
Effect on Eating Disorder Symptomatology (multiple variables) 8. sleep quality | 1 year
  Consensus Sleep Diary (CSD). 15 items to prospectively assess subjective estimates of daily sleep patterns, including time eyes closed, sleep-onset latency, number of awakenings, time of final awakening, and total time spent awake after sleep onset. Additional items include a Likert rating of sleep quality, medication use, and naps.Sleep diaries are universally the preferred method for collecting self-reported sleep data. There is no score on this measure Patient-Reported Outcomes Measurement Information System (PROMIS) Pediatric Sleep Disturbance and Sleep-Related Impairment, 8-item short forms. The PROMIS Pediatric Sleep Disturbance and Sleep-Related Impairment item banks are self-report eight item measures that assesses perceptions of sleep depth, restoration, and quality over the past seven days. Higher scores indicating greater sleep/wake disturbances.
Effect on Eating Disorder Symptomatology (multiple variables) - 9. expressed emotion | 1 year
  Expressed Emotion measured by Difficulties in Emotional Regulation (DERS). The DERS is a self-report measure of subjective emotion ability, as defined by a prominent clinically derived model of emotion regulation. Higher scores suggest greater problems with emotion regulation.
Effect on Eating Disorder Symptomatology (multiple variables) - 10. expressed emotion | 1 year
  Expressed Emotion measured by Brief Dyadic Scale of Expressed Emotion This is a 14 item self-report questionnaire. The items of this self- report measure are scored on a 10-point Likert scale. Higher scores indicate higher levels of criticism/expressed emotion.
Effect on Eating Disorder Symptomatology (multiple variables) - 11. expressed emotion | 1 year
  Expressed Emotion measured by Family Questionnaire (FQ) The Family Questionnaire (FQ),is The Family Questionnaire (FQ) is a 20-item, self-administered questionnaire that measures expressed emotion status (criticism and emotional over involvement [EOI]) of family members toward patients with mental illness. Expressed Emotion measured by Family Questionnaire (FQ) The FQ has two sub-scales: critical comments, and EOI. Each item is rated on a 4-point scale (1 = never/very rarely; 4 = very often). The FQ is scored by adding together the ratings from the individual items, with higher scores indicating greater levels of expressed emotion.
Effect on Eating Disorder Symptomatology (multiple variables) - 12. Parenting styles | 1 year
  Parenting Styles categorized by Diana Baumrind's 4 parenting styles including authoritative, authoritarian, permissive, and uninvolved parenting styles. This is assessed by the MFT intensive leaders at the beginning of the MFT intervention at Day 1 and then again at Day 4. This assessment results in parents being categorized into one of the 4 parenting styles.

SECONDARY OUTCOMES:
Implementation and feasibility of virtual adaptation of MFT 1. participant retention | 4 years
  evaluate participant retention - This is calculating drop out scores as a percentage of total participants.
Implementation and feasibility of virtual adaptation of MFT - 2. participant satisfaction | 4 years
  Participant satisfaction of program measured by MFT Feedback Form (created by investigators).This is a qualitative measure seeking subjective responses from participants related to their overall experience in the program.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No